CLINICAL TRIAL: NCT05036382
Title: A Study on Analysis of Factors to Affect the Provision of Health Data of Users Through the Personal Health Management Application
Brief Title: Factors to Affect the Provision of Health Data of Users Through PHR App
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: clinical trials_1
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-06

CONDITIONS: Personal Health Record
Keywords: PHR; Incentive Mechanism; Token Economy; Data Sharing; Lifelog data; RCT; Personal Health Record; Health Mobile app

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: A group that receives an incentive message one month after the start of the experiment
  Interventions: Behavioral: Steps data observation
- Control Group: A group that does not receive an incentive message (for equity, incentive messages will be sent in the last month of the experiment)

INTERVENTIONS:
Behavioral: Steps data observation — Sending more step data from the experimental group that received the incentive message
  Groups: Experimental Group

SUMMARY:
An experiment to determine if the incentive message affects people's active health data sharing.

DETAILED DESCRIPTION:
Researchers send a weekly message to participants asking them to share their step data on their personal health records(PHR) applications. (4months in total)

(Baseline, 1month) For the first month, researchers send the same data request message to both counties.

1. term, 1 month) The researchers added a message saying, 'Incentives are provided for data sharing' only to the experimental group.
2. term, 1 month) Excludes incentive message for both groups
3. term, 1 month) The researchers added a message saying, 'Incentives are provided for data sharing' only to the control group.

   * For equity in both groups, an incentive message was provided to the control group in the last month under the same conditions as the experimental group.
   * Only the first 3 months of data were used for the study.

Hypothesis

* In 1-term, the number of data sharing in the experimental group is higher than that in the control group.
* In 1-term, the number of data sharing in the experimental group is more active than baseline period.
* In 2-term, the number of data sharing in the experimental group is still higher than in the baseline period.
* Over the next 1 month, the number of sharing in the experimental group was maintained, which was still higher than that of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 to 70
* A person who has no difficulty in installing and using PHR app under study
* A person who has expressed his/her willingness to participate voluntarily

Exclusion Criteria:

* Children/Adolescents under the age of 18 or Seniors over 71 years of age
* Those who do not have a smartphone or who are not proficient in using a smartphone
* Persons who are uncooperative and difficult to understand the research method due to cognitive decline

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with smartphones that have no problems installing and using health applications
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-25 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Average number of data shares | 3 months
  The average number of steps data sharing between the experimental group and the control group according to the incentive message

SECONDARY OUTCOMES:
Percentage of participants with increased number of shares compared to baseline-term | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Gyeonggi-do, Bundang-gu, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: No